CLINICAL TRIAL: NCT02848508
Title: Metformin in Moderate and Severe Renal Failure (CKD 3-4): A Follow-up Study
Acronym: METsuiviIRC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2016_843_0009
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Metformin; moderate renal failure; severe renal failure; chronic kidney disease; hyperlactatemia; lactic acidosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Hyperlactatemia; Acidosis, Lactic | interventions — Metformin

ARMS (3):
- moderate impairment, CKD stage 3a (Experimental): (12 subjects): GFR 59-45 (moderate impairment, CKD stage 3a) Metformin : 1500mg/day
  Interventions: Drug: Metformin
- moderate impairment, CKD stage 3a) (Experimental): (12subjects): GFR 44-30 (moderate impairment, CKD stage 3b) Metformin : 1000mg/day
  Interventions: Drug: Metformin
- severe impairment (Experimental): (12 subjects): GFR 29-15 (severe impairment, CKD stage 4) Metformin : 500mg/day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin
  Other Names: Glucophage

SUMMARY:
To validate on the mid-term in moderate and severe renal failure (CKD 3-4) a nomogram to adapt a fixed metformin daily posology according to renal function on the basis of the first short-term study made by the investigators.

DETAILED DESCRIPTION:
A first open-label pilot study at different stages of CKD (1-5) (concerning whether or not metformin use is safe provided a dose adjustment is used) has evaluated (i) metformin levels in plasma and in erythrocytes according to an increasing metformin dosage and CKD severity (1-5) and (ii) the prevalence of lactate levels ≥2.5 mmol/L in CKD 3-5. All patients underwent 3 one-week- blocks of metformin treatment at an increasing dosage, each of which followed by a one week-wash- out period: 500 mg/day in the evening (E) in phase 1; 1,000 mg/day (500 mg morning (M) and E) in phase 2; 2,000 mg/day (1,000 mg M and E) in phase 3.

Steady-state trough blood levels were assayed 12 hours after the last dose of metformin. In this study a progressive dose-related increase of the trough metformin levels were observed and in particular in severe CKD stages. No case of severe hyperlactatemia was reported in this study. In continue, the investigators thought to conduct a new study to evaluate safety of metformin in mid-term period of time. For this purpose, metformin will be given at a fixed dose during 4 months: 1) 1,500 mg/day (500 mg M and 1,000 mg E) in stage 3a; 2) 1,000 mg/day (500 mg M and E) in stage 3b; and 3) 500 mg/day (M) in stage 4. Metformin levels in plasma and in erythrocytes, venous lactate, and HbA1c levels will be measured at 1, 2, 3 and 4 months for assessment of safety.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients with stable CKD stages 3A, 3B and 4 aged between 18 and 80 years requiring metformin (and any other antidiabetic treatment)

Exclusion Criteria:

* Hyperlactatemia (> 2.5 mmol/L)
* No creatinine levels available since 3 months
* Severe hepatic insufficiency
* No liver function parameters available
* Need of investigation with iodized contrast media
* Hypersensitivity to metformin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Monitoring of blood metformin plasma levels with a fixed dose of metformin | 4 months
Monitoring of blood metformin erythrocytes levels with a fixed dose of metformin | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Daniel LALAU, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France